CLINICAL TRIAL: NCT00600769
Title: Open Study of Clarithromycin for the Treatment of Infections Caused by Nontuberculous Mycobacteria (NTM)
Brief Title: Clarithromycin for the Treatment of Infections Caused by Nontuberculous Mycobacteria (NTM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Richard J. Wallace, Jr., M.D., Chairman Department of Microbiology, The University of Texas Health Science Center at Tyler
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 263
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Nontuberculous Mycobacteria; Mycobacterium Avium Complex
Keywords: MAC; NTM
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection | interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment of MAC and other NTM (Other): Clarithromycin drug given twice daily.
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin — Dosage dependent on clinical factors such as age, weight and patient-specific health status
  Other Names: Biaxin

SUMMARY:
Use of oral clarithromycin for treatment of chronic lung disease due to Mycobacterium avium-intracellulare and other non-tuberculous Mycobacteria

DETAILED DESCRIPTION:
Oral clarithromycin for treatment of MAC and other nontuberculous mycobacteria in adults with clinical history

ELIGIBILITY:
Inclusion Criteria:

* Meet American Thoracic Society criteria for nontuberculous lung disease: two or more AFB smear positive, culture positive sputums or bronchoscopic samples and/or two or more AFB smear negative respiratory samples with moderate to heavy growth (2+-4+); abnormal CXR consistent with M. avium lung disease; absence of other potential lung pathogens (except for the coexistence of M. abscessus)
* Age 18 years and older

Exclusion Criteria:

* History of macrolide allergy
* Must not receive the antihistamines terfenadine (Seldane) or astemizole (Hismanal) while on clarithromycin
* Children less than 18 years of age
* If a menstruating female, not pregnant and on adequate birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 1991-01 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Clinical and microbiological outcomes, such as clinical symptoms and laboratory cultures | 6 months
  neg culture x3( sputum conversion)

SECONDARY OUTCOMES:
Microbiological cultures | 1yr
  neg culture for 1 yr on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Wallace, MD, Principal Investigator — UTHSCT
Locations (1):
- The University of Texas Health Science Center at Tyler, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No